CLINICAL TRIAL: NCT03826940
Title: Linking Inhibition From Molecular to Systems and Cognitive Levels: a Preclinical and Clinical Approach in Autism Spectrum Disorders and Neurofibromatosis.
Brief Title: From Molecules to Cognition: Inhibitory Mechanisms in ASD and NF1
Acronym: ASD/NF1inhib
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Miguel Castelo-Branco, Research Director of CIBIT-ICNAS, University of Coimbra
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CRU2C-ICNAS-001; FLAD Life Science 2020 (Other Grant/Funding Number: Luso-American Development Foundation)
Record Dates: First submitted 2019-01-23; First posted 2019-02-01 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2020-11

CONDITIONS: Autism Spectrum Disorder; Neurofibromatosis 1
Keywords: Inhibition; GABA; molecular imaging; functional magnetic resonance imaging; Autism Spectrum Disorder; Neurofibromatosis 1
MeSH Terms: conditions — Autism Spectrum Disorder; Neurofibromatosis 1; Inhibition, Psychological | interventions — Lovastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- NF1 - experimental (Experimental)
  Interventions: Drug: Lovastatin 60 MG
- NF1 - control (Placebo Comparator)
  Interventions: Drug: Placebos
- ASD - experimental (Experimental)
  Interventions: Drug: Lovastatin 60 MG
- ASD - control (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Lovastatin 60 MG — 60 MG Lovastatin per day for 3 consecutive days
  Arms: ASD - experimental; NF1 - experimental
Drug: Placebos — 60 MG Placebo per day for 3 consecutive days
  Arms: ASD - control; NF1 - control

SUMMARY:
This study aims to investigate synaptic physiology and behavioral inhibition in patients with NF1 and ASD and to answer whether inhibitory deficits at these levels are modulated by lovastatin.

Structure: (1) Visit 1: Baseline assessment- participant's characterization, baseline outcome measures and additional evaluations, (2) 3 consecutive days of physiologically probing drug/placebo intake, (3) Visit 2: Outcome measures and additional evaluations in the day after the last drug/placebo intake, (4) Washout period of 4 to 6 weeks, (5) 3 consecutive days of drug/placebo intake, (6) Visit 3: Outcome measures and additional evaluations in the day after the last placebo/drug intake.

DETAILED DESCRIPTION:
The literature has shown synaptic inhibitory dysfunction in both ASD and NF1. Here the investigators aim to test whether a mechanistic link can be established between that synaptic inhibitory dysfunction, systems levels changes in oscillatory synchrony and regulation of inhibition and treatment with Lovastatin in these two neurodevelopmental disorders. The investigators will explore this link through the application of complementary quantitative measures (putative biomarkers), such as magnetic resonance spectroscopy (MRS) transcranial magnetic stimulation (TMS) and electroencephalogram (EEG) applied to the same group of adult patients before and after the lovastatin or placebo intake during three days.

The intervention comprehends three sessions: the first two visits will occur in the same week and the third visit will take place 4 to 6 weeks later. In the first visit (baseline assessment), participants will perform neuropsychological, EEG, MRS and TMS assessment. In the other two visits participants will repeat EEG, MRS and TMS assessments to study possible post- intervention effects. Participants will intake 60mg of Lovastatin or Placebo during three consecutive days before the second and the third visits.

ELIGIBILITY:
Inclusion Criteria:

* Positive diagnostic results for ASD in:

The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria.

* Positive diagnostic results for NF1:

Clinical diagnosis based on the well-established clinical criteria

Exclusion Criteria:

* Global Intelligence Quotient < 80
* Associated medical condition such as epilepsy, neurologic conditions, genetic syndromes, or other usual comorbidity in ASD and NF1 populations
* Medication capable of interfering with the intervention and/or study results
* Pregnancy
* Drug use and/or alcohol abuse
* Contra-indications to MR and TMS

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Neurochemical response changes to GABAergic stimulation | Through study completion, an average of 1 year
  Comparing changes in brain excitation-inhibition measures (i.e., glutamate and GABA) when the GABAergic system is activated by oral dose of the Lovastatin 60mg during 3 days versus the placebo condition.

SECONDARY OUTCOMES:
Motor evoked potentials changes under motor cortical stimulation | Through study completion, an average of 1 year
  Amplitudes (mV) will be measured during stimulation of the primary motor cortex using transcranial magnetic stimulation
Cortical excitability changes under motor cortical stimulation | Through study completion, an average of 1 year
  Periods (ms) will be measured during stimulation of the primary motor cortex using transcranial magnetic stimulation
Brain oscillations changes under sensory stimulation | Through study completion, an average of 1 year
  Power (microV^2) will be recorded during sensory stimulation using high density electroencephalography.
Event-related potentials changes under sensory stimulation | Through study completion, an average of 1 year
  Amplitude (microV) will be recorded during sensory stimulation using high density electroencephalography.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel S Castelo-Branco, MD, PhD, Principal Investigator — ICNAS - Institute of Nuclear Sciences Applied to Health
Locations (1):
- ICNAS, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pizzarelli R, Cherubini E. Alterations of GABAergic signaling in autism spectrum disorders. Neural Plast. 2011;2011:297153. doi: 10.1155/2011/297153. Epub 2011 Jun 23. PMID 21766041
- [Background] Violante IR, Ribeiro MJ, Edden RA, Guimaraes P, Bernardino I, Rebola J, Cunha G, Silva E, Castelo-Branco M. GABA deficit in the visual cortex of patients with neurofibromatosis type 1: genotype-phenotype correlations and functional impact. Brain. 2013 Mar;136(Pt 3):918-25. doi: 10.1093/brain/aws368. Epub 2013 Feb 11. PMID 23404336
- [Derived] Bernardino I, Dionisio A, Castelo-Branco M. Cortical inhibition in neurofibromatosis type 1 is modulated by lovastatin, as demonstrated by a randomized, triple-blind, placebo-controlled clinical trial. Sci Rep. 2022 Aug 15;12(1):13814. doi: 10.1038/s41598-022-17873-x. PMID 35970940